CLINICAL TRIAL: NCT02842749
Title: Phase IV, Open-label, Multi-center, Single-arm Study of the Safety and Efficacy of Everolimus (Afinitor) in Adult Patients With Locally Advanced, Unresectable or Metastatic, Well Differentiated Progressive Pancreatic Neuroendocrine Tumors (pNET) in China.
Brief Title: Phase IV Study of the Safety and Efficacy of Everolimus in Adult Patients With Progressive pNET in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001PCN31
Record Dates: First submitted 2016-06-16; First posted 2016-07-25 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Neuroendocrine Tumors
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- everolimus (single arm) (Experimental): Participants were instructed to take everolimus at a starting dose of 10 mg orally once daily. However, dose adjustments were permitted in order to allow the participant to continue the study treatment.
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — Participants were instructed to take everolimus at a starting dose of 10 mg orally once daily. However, dose adjustments were permitted in order to allow the participant to continue the study treatment.

SUMMARY:
To evaluate safety and efficacy of everolimus (Afinitor®) in Chinese adult patients with local advanced or metastatic, well differentiated progressive pancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
This was an open-label, multicenter, single-arm clinical study to evaluate the safety and efficacy of everolimus in Chinese adult patients with locally advanced, unresectable or metastatic, well differentiated progressive pancreatic neuroendocrine tumors. The inclusion and exclusion criteria, as well as the dosing and dose modification criteria are designed according to the approved Chinese Package Insert. The planned sample size of the study was approximately 60 subjects.

Subjects who were eligible received the treatment with everolimus provided by sponsor to treat pNET and followed the visit schedule in the protocol to collect safety and efficacy data until progression of disease, unacceptable toxicity, death, protocol deviation or other reason that may lead to discontinuation before the end of study. All subjects were followed-up for survival status every 6 months by the investigator until death, lost to follow-up, withdrawal of consent for survival or end of study.

The "End of study" is defined as either at least 75% of subjects have completed survival follow up or all subjects discontinued study treatment or the last subject finished 5-year survival follow up, whichever comes first. Final analysis was conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmed G1 or G2 pancreatic neuroendocrine tumors(pNETs) (WHO 2010)
* Patients must have radiological documentation of progression of disease per RECIST 1.1 within 12 months prior to enrollment.
* Measurable disease per RECIST 1.1 criteria using triphasic computed tomography (CT) scan or multiphase MRI for radiologic assessment.
* everolimus treatment which is recommended by the treating physician

Exclusion Criteria:

* Hypersensitivity to everolimus, to other rapamycin derivatives, or to any of the excipients.
* Patient who is unwilling to receive Afinitor treatment due to any reason.
* Pregnant or nursing (lactating) women,
* Prior therapy with mTOR inhibitors (e.g. sirolimus, temsirolimus, everolimus).
* Use of an investigational drug within the 30 days prior to enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- China (4):
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 5 investigative sites in China.
Period: Overall Study
Arm/Group | Everolimus
Started | 61
Completed | 61
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.22 (14.305)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with treatment emergent adverse events (any AE regardless of seriousness), SAEs, AEs and SAEs on grade 3 or 4, and suspected to be related to the study drug.
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period of 30 days, up to a maximum duration of approximately 5 years.
Population: Safety Analysis Set (SS): including all participants who received at least one study treatment. Participants were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 61
Participants
  AEs | 60
  AEs-grade 3/4 | 30
  AEs Suspected to be related to the study drug | 58
  AEs Suspected to be related to the study drug-grade 3/4 | 19
  SAEs | 17
  SAEs-grade 3/4 | 11
  SAEs Suspected to be related to the study drug | 8
  SAEs Suspected to be related to the study drug-grade 3/4 | 5

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from the start of study treatment to death due to any cause. OS was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 7 years and 6 months.
Population: Full Analysis Set (FAS): including all participants who received at least one study treatment. Participants were analyzed according to the treatment they actually received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 61
months | 66.56 [39.66 to NA] — Not estimable due to insufficient number of participants with events

3. Secondary Outcome: Progression Free Survival (PFS) by Investigator Assessment Per RECIST 1.1
Description: Progression free survival is defined as the time from the initiation of study treatment to disease progression or death due to any cause. PFS was analyzed using Kaplan-Meier estimates.
Time Frame: Up to approximately 2 years and 9 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 61
months | 16.07 [11.04 to 21.52]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days (on treatment period), up to a maximum duration of approximately 5 years. All cause mortality was reported until end of study, up to approximately 7 years and 6 months (on treatment plus survival follow-up period).
Description: Adverse events were only collected in the on treatment period. Deaths in the post treatment survival follow up period are not considered AEs.
Groups:
- Everolimus-on Treatment: AEs collected from randomization up to 30 days post-treatment
- Everolimus-Survival Follow-up: Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Everolimus-on Treatment | Everolimus-Survival Follow-up
All-Cause Mortality (participants affected / at risk) | 6/61 | 22/55
Serious Adverse Events (participants affected / at risk) | 17/61 | 0/0
Other Adverse Events (participants affected / at risk) | 60/61 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus-on Treatment (N=61) | Everolimus-Survival Follow-up (N=0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | NA
Cachexia (Metabolism and nutrition disorders) | 1 | NA
Function liver abnormal (Hepatobiliary disorders) | 1 | NA
Infectious pneumonitis (Infections and infestations) | 3 | NA
Anal abscess (Infections and infestations) | 1 | NA
Sepsis (Infections and infestations) | 1 | NA
Herpes virus infection (Infections and infestations) | 1 | NA
Hemorrhage cerebral (Nervous system disorders) | 1 | NA
Hypoglycemic encephalopathy (Nervous system disorders) | 1 | NA
Hepatic encephalopathy (Nervous system disorders) | 1 | NA
Movement disorder (Nervous system disorders) | 1 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Tumor rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Asthenia (General disorders) | 2 | NA
Fever (General disorders) | 1 | NA
Death (General disorders) | 1 | NA
Renal failure (Renal and urinary disorders) | 1 | NA
Vomiting (Gastrointestinal disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus-on Treatment (N=61) | Everolimus-Survival Follow-up (N=0)
Hypokalaemia (Metabolism and nutrition disorders) | 11 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 7 | NA
Decreased appetite (Metabolism and nutrition disorders) | 7 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 5 | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | NA
Upper respiratory tract infection (Infections and infestations) | 4 | NA
Aspartate aminotransferase increased (Investigations) | 27 | NA
Alanine aminotransferase increased (Investigations) | 18 | NA
White blood cell count decreased (Investigations) | 16 | NA
Neutrophil count decreased (Investigations) | 15 | NA
Platelet count decreased (Investigations) | 14 | NA
Blood glucose increased (Investigations) | 13 | NA
Weight decreased (Investigations) | 9 | NA
Blood alkaline phosphatase increased (Investigations) | 9 | NA
Gamma-glutamyltransferase increased (Investigations) | 7 | NA
Blood albumin decreased (Investigations) | 7 | NA
White blood cell count increased (Investigations) | 6 | NA
Lymphocyte count decreased (Investigations) | 6 | NA
Blood cholesterol increased (Investigations) | 6 | NA
Blood lactate dehydrogenase increased (Investigations) | 6 | NA
Low density lipoprotein increased (Investigations) | 5 | NA
Haemoglobin decreased (Investigations) | 5 | NA
Neutrophil count increased (Investigations) | 5 | NA
Activated partial thromboplastin time prolonged (Investigations) | 4 | NA
Protein urine present (Investigations) | 4 | NA
Blood bilirubin increased (Investigations) | 4 | NA
Blood triglycerides increased (Investigations) | 4 | NA
Blood creatinine increased (Investigations) | 4 | NA
Infectious pneumonitis (Infections and infestations) | 6 | NA
Headache (Nervous system disorders) | 4 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | NA
Rash (Skin and subcutaneous tissue disorders) | 15 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 6 | NA
Pyrexia (General disorders) | 13 | NA
Oedema peripheral (General disorders) | 13 | NA
Asthenia (General disorders) | 13 | NA
Proteinuria (Renal and urinary disorders) | 9 | NA
Mouth ulceration (Gastrointestinal disorders) | 24 | NA
Stomatitis (Gastrointestinal disorders) | 23 | NA
Diarrhoea (Gastrointestinal disorders) | 22 | NA
Abdominal discomfort (Gastrointestinal disorders) | 5 | NA
Vomiting (Gastrointestinal disorders) | 5 | NA
Abdominal pain (Gastrointestinal disorders) | 4 | NA
Abdominal distension (Gastrointestinal disorders) | 4 | NA
Hypertension (Vascular disorders) | 9 | NA
Anaemia (Blood and lymphatic system disorders) | 30 | NA
Eyelid oedema (Eye disorders) | 4 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT02842749/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT02842749/SAP_001.pdf